CLINICAL TRIAL: NCT02795208
Title: Lung Recruitment Improves Right Ventricle Performance After Cardio-Pulmonary Bypass
Brief Title: Lung Recruitment Improves Right Ventricle Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Privado de Cordoba, Argentina (Other)
Responsible Party: Principal Investigator, Silvina Longo, Medical Doctor, Hospital Privado de Cordoba, Argentina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HPrivadoCordoba
Record Dates: First submitted 2016-06-05; First posted 2016-06-10 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Atelectasis
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Patients received standard protective ventilation along the protocol.
- Recruitment maneuver group (Experimental): Patient received a lung recruitment maneuver after cardiopulmonary bypass. The recruitment maneuver consists in 10 breaths at 40/20 cmH2O of plateau pressure and PEEP, respectively. Then, the .ventilatory settings back to protective ventilation but adding 10 cmH2O of PEEP to keep the lungs open.
  Interventions: Procedure: Lung recruitment maneuver

INTERVENTIONS:
Procedure: Lung recruitment maneuver — The lung recruitment maneuver consists in a brief and controlled increment in airways pressure (20 cmH2O of PEEP + 20 cmH2O of driving pressure) for 10 breaths.
  Arms: Recruitment maneuver group

SUMMARY:
This study test whether a lung recruitment maneuver improves the right ventricle performance after cardiopulmonary bypass. Half of the patients received an standard protective ventilation and the other half the same ventilatory pattern after a lung recruitment maneuver.

DETAILED DESCRIPTION:
Atelectasis is developed in 90% of anesthetized patients after surgery.

Protective ventilation with low tidal volumes and positive-end expiratory pressure (PEEP) promotes atelectasis with the potential right ventricle dysfunction induced by the increment in afterload (activation of the pulmonary hypoxic vasocontriction reflex).

Lung recruitment can improve the right ventricle performance caused by atelectasis because the pulmonary hypoxic vasocontriction reflex desapear in a normal aerated lungs.

ELIGIBILITY:
Inclusion Criteria:

* cardiovascular surgery with cardiopulmonary bypass.
* Patients with a New York Heart Association (NYHA) class I-II,
* Pre-operative left ventricular ejection fraction ≥ 50 %.
* Euroscore ≤ 6.

Exclusion Criteria:

* TEE contraindications.
* Hemodynamically unstable
* Needi for inotropic support

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-03; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Right ventricle assessment by transesophageal echocardiography | intraoperative

SECONDARY OUTCOMES:
Atelectasis assessment by transesophageal echocardiography | intraoperative
PaO2 and respiratory compliance | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Silvina Longo, MD, Principal Investigator — Hospital Privado de Córdoba

IPD SHARING:
Plan to Share IPD: Undecided